CLINICAL TRIAL: NCT02853396
Title: A Pilot of a Brief Cognitive Behaviour Therapy Formulation Focused Intervention for Internalised Stigma With Acute Inpatients That Experience Psychosis
Brief Title: A Study of an Cognitive Behaviour Therapy for Internalised Stigma Intervention for Inpatients With Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lisa Wood (Other)
Responsible Party: Sponsor-Investigator, Lisa Wood, Clinical Psychologist, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/NW/0332
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Cognitive Behaviour Therapy for Internalised Stigma; Psychoeducation
Keywords: internalised stigma; self stigma; inpatients; CBT; Cognitive therapy
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioural therapy (Experimental): Cognitive behaviour therapy
  Interventions: Other: Cognitive Behaviour Therapy
- Psychoeducation (Active Comparator): psychoeducation
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Other: Cognitive Behaviour Therapy
  Arms: Cognitive behavioural therapy
Other: Psychoeducation
  Arms: Psychoeducation

SUMMARY:
Stigma is a significant concern for those who experience psychosis. People with psychosis are the most stigmatised group of all mental health difficulties. There is a lack of research examining the effectiveness of psychological therapies for people who experience psychosis who are also experiencing negative impacts of stigma. To date, all studies examining stigma therapies have been conducted with outpatients and no support have been developed for inpatients. The aim of this study to conduct a pilot randomised controlled trial of a brief therapy (based on cognitive behavioural therapy)to help participants cope with stigma. It will be compared to a educational control intervention. Both therapies will last approximately two hours and be conducted in one or two sessions by the principal investigator (clinical psychologist). Participants will be given a number of questionnaires assessing a number of outcomes such as impacts of stigma, depression, recovery, and self-esteem. Participants will be assessed on these measure prior to the therapy, post therapy and at follow-up.

DETAILED DESCRIPTION:
A single-blind randomised controlled pilot trial will be conducted comparing a Cognitive Behaviour Therapy formulation driven internalised stigma intervention (experimental group) against a psychoeducational control intervention (control group). It will follow recommendations outlined by the Medical Research Council's framework for the development and evaluation of complex interventions. This will allow for the medication of the intervention if necessary in order to examine what type of intervention is best suited to the inpatient environment.

Aim: To examine the efficacy of a formulation driven intervention for internalised stigma in psychosis with acute inpatients. The intervention will be compared to a brief psychoeducational internalised stigma intervention.

Description of therapies:

Experimental Condition The experimental condition will receive a two hour intervention session (across one or two sessions) which will be based on a Cognitive Behaviour therapy formulation. These sessions will be undertaken within a two week period. The sessions will collaboratively assess and create a narrative of the participants' experiences of stigma, and develop a personalised stigma formulation. A stigma-related goal will be identified and a brief intervention will be collaboratively developed to tackle this goal. The intervention formulation and change mechanisms will draw upon strategies for people who experience psychosis. Intervention strategies may include guided discovery, skills development, normalising and belief change strategies, including behavioural experiments targeting stigma-relevant appraisals and negative beliefs about self including public stereotypes of psychosis, and supporting decisions about whether to disclose.

Control Condition The control condition will receive a two hour session receiving psychoeducation and normalising material relating to stigma in psychosis. The aim of the material is normalise experiences of psychosis and stigma. Information includes prevalence rates of psychosis, experiences of stigma and discrimination commonly reported by those who experience psychosis.

Both interventions will be delivered by the same therapist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65
* Who meet criteria for a schizophrenia-spectrum diagnoses (schizophrenia, schizophreniform disorder, schizoaffective disorder, delusional disorder or psychotic disorder not otherwise specified; ICD-10)
* Able to give in-formed consent and have capacity to consent
* Receiving care from a clinical in-patient team
* Able to complete the interview in English
* Self-report being concerned about stigma

Exclusion Criteria:

* Non-English speakers (due to translation costs)
* An acquired brain injury or substance misuse judged to be the acute cause of the psychotic experiences
* Lacking capacity for informed consent (the applicant will work with the participant to assess whether they understand the information sheet and study and therefore their ability to give informed consent)
* Experiencing severe thought disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-02 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Internalised stigma of mental illness scale | 10 minutes

SECONDARY OUTCOMES:
Process of Recovery Questionnaire | 5 minutes
Beck Depression Inventory | 5 minutes
Beck Hopelessness Scale | 5 mins
Self-Esteem Rating scale | 5 mins
Attitudes towards mental health scale | 5 mins

CONTACTS AND LOCATIONS:
Locations (1):
- North east london foundation trust, Ilford, Essex, United Kingdom

REFERENCES:
- [Derived] Wood L, Byrne R, Enache G, Morrison AP. A brief cognitive therapy intervention for internalised stigma in acute inpatients who experience psychosis: A feasibility randomised controlled trial. Psychiatry Res. 2018 Apr;262:303-310. doi: 10.1016/j.psychres.2017.12.030. Epub 2017 Dec 13. PMID 29494866